CLINICAL TRIAL: NCT04706325
Title: INVESTIGATION OF RISK FACTORS RELATED TO COVID-19 RELATED KIDNEY DAMAGE: A PROSPECTIVE OBSERVATIONAL STUDY
Brief Title: COVID-19 RELATED KIDNEY DAMAGE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kocaeli Derince Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Aki̇f Şahi̇n, md, Kocaeli Derince Education and Research Hospital
Other Study IDs: kocaeli derh
Record Dates: First submitted 2021-01-11; First posted 2021-01-12 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- COVİD19 PCR (Polymerase Chain Reaction) AND CT POSITIVE: COVİD19 PCR (Polymerase Chain Reaction) AND CT POSITIVE
  Interventions: Other: ACUTE KIDNEY INJURY
- COVİD19 PCR (Polymerase Chain Reaction)NEGATİVE AND CT POSITIVE: COVİD19 PCR (Polymerase Chain Reaction)NEGATİVE AND CT POSITIVE
  Interventions: Other: ACUTE KIDNEY INJURY
- COVİD19 PCR (Polymerase Chain Reaction) AND CT will be evaluated as NEGATIVE.: COVİD19 PCR (Polymerase Chain Reaction) AND CT will be evaluated as NEGATIVE.
  Interventions: Other: ACUTE KIDNEY INJURY

INTERVENTIONS:
Other: ACUTE KIDNEY INJURY — KDIGO LEVELS

SUMMARY:
In this study, we investigate whether the early detection of risk factors in Covid-19 associated acute kidney injury contributes to us in the early initiation of treatment. We predict that if acute kidney damage is detected early in patients with early risk factors, permanent kidney damage will be seen less. In addition, we think that covid-19 patients may have positive contributions to shortening treatment time and reducing treatment costs. In addition, we are investigating whether it has a positive effect on patients' survival. In other words, we are investigating the contribution of risk factors to early diagnosis and treatment, the effect on health expenditures and mortality in patients with COVID-19 with acute kidney damage.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 aged
* patients in ICU

Exclusion Criteria:

* Patients with known Chronic Renal Failure
* who have received dialysis treatment before
* who are under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Over 18 aged
  * patients in ICU
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-05-15 (Estimated)

PRIMARY OUTCOMES:
KDIGO | 4 MONTHS
  Kidney Disease: Improving Global Outcomes

CONTACTS AND LOCATIONS:
Overall Officials: akif şahin, Principal Investigator — kocaeli derh
Locations (1):
- Akif Şahin, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cheng Y, Luo R, Wang K, Zhang M, Wang Z, Dong L, Li J, Yao Y, Ge S, Xu G. Kidney disease is associated with in-hospital death of patients with COVID-19. Kidney Int. 2020 May;97(5):829-838. doi: 10.1016/j.kint.2020.03.005. Epub 2020 Mar 20. PMID 32247631
- [Result] Aleebrahim-Dehkordi E, Reyhanian A, Saberianpour Sh, Hasanpour-Dehkordi A. Acute kidney injury in COVID-19; a review on current knowledge. J Nephropathol. 2020;9:e31. doi: 10.34172/jnp.2020.31
- [Result] Alhazzani W, Moller MH, Arabi YM, Loeb M, Gong MN, Fan E, Oczkowski S, Levy MM, Derde L, Dzierba A, Du B, Aboodi M, Wunsch H, Cecconi M, Koh Y, Chertow DS, Maitland K, Alshamsi F, Belley-Cote E, Greco M, Laundy M, Morgan JS, Kesecioglu J, McGeer A, Mermel L, Mammen MJ, Alexander PE, Arrington A, Centofanti JE, Citerio G, Baw B, Memish ZA, Hammond N, Hayden FG, Evans L, Rhodes A. Surviving Sepsis Campaign: guidelines on the management of critically ill adults with Coronavirus Disease 2019 (COVID-19). Intensive Care Med. 2020 May;46(5):854-887. doi: 10.1007/s00134-020-06022-5. Epub 2020 Mar 28. PMID 32222812